CLINICAL TRIAL: NCT03252106
Title: Long-term Effectiveness of Contour Augmentation in Sites With Early Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P004 Study
Record Dates: First submitted 2017-07-19; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Jaw, Edentulous, Partially; Dental Implants, Single-tooth; Grafting Bone
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contour augmentation (Experimental)
  Interventions: Procedure: Contour augmentation with implant placement

INTERVENTIONS:
Procedure: Contour augmentation with implant placement — Contour augmentation with implant placement

SUMMARY:
In this prospective case series study, 20 patients with an implant-borne single crown following early implant placement with simultaneous contour augmentation will be followed for 10 years. Clinical, radiologic, and esthetic parameters will be assessed. In addition, cone beam computed tomography (CBCT) will be used at 10 years to examine the facial bone wall and compared to the 6 year data.

ELIGIBILITY:
Inclusion Criteria:

* Single tooth gaps post extraction in the esthetic zone
* Written informed consent

Exclusion Criteria:

* Heavy smoking (more than 10 cigarettes per day)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-11-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness of contour augmentation | 10 year examination
  Measurement of facial bone wall width with cone beam CTs (in mm)

SECONDARY OUTCOMES:
Esthetic examination | 10 year examination
  Pink Esthetic Score
Peri-Implant soft tissue health | 10 year examination
  Plaque Index
Peri-implant bone loss over time | 10 year examination
  Distance from the implant-shoulder to the first bone-to-implant-contact (DIB) in mm
Peri-Implant soft tissue health | 10 year examination
  Sulcus Bleeding Index

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Buser, DMD, Study Chair — University of Bern
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Chappuis V, Rahman L, Buser R, Janner SFM, Belser UC, Buser D. Effectiveness of Contour Augmentation with Guided Bone Regeneration: 10-Year Results. J Dent Res. 2018 Mar;97(3):266-274. doi: 10.1177/0022034517737755. Epub 2017 Oct 26. PMID 29073362